CLINICAL TRIAL: NCT05753956
Title: A Phase 1 Clinical Trial to Determine the Safety, Pharmacokinetics and Pharmacodynamics of Intravenous GH002 in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of GH002 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GH Research Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GH002-HV-105; 2022-002620-13 (EudraCT Number)
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
Keywords: 5-MeO-DMT; 5-methoxy-N,N-dimethyltryptamine; Healthy Volunteers; Pharmacokinetics; Mebufotenin
MeSH Terms: interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Intervention Model Description: This study will include separate single and multiple-dose parts.
  Single-dose Part:
  A double-blind, placebo-controlled, randomized, dose escalation design with single doses of GH002 delivered by i.v. bolus injection in 7 consecutive cohorts with 8 subjects per cohort (randomized as 6 active and 2 placebo):
  Cohort A: Dose A
  Cohort B: Dose B
  Cohort C: Dose C
  Cohort D: Dose D
  Cohort E: Dose E
  Cohort F: Dose F
  Cohort G: Dose G
  Up to 2 additional cohorts may be added before the IDR part is initiated. These will be named cohorts H and I, if needed.
  Multiple-Dose Part:
  An open-label, non-randomized design with up to 3 doses of GH002 administered to subjects by i.v. bolus injection(s) on a single day in one cohort of 8 subjects:
  Cohort J: Individualized Dosing Regimen with GH002.
  The exact doses of study drug to be administered will be determined after an unblinded review of the safety, PK and PD data from all of the cohorts in the single dose part of the trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort A: Dose A single dose (Experimental): A single dose of GH002 or placebo administered by i.v. bolus injection (randomized as 6 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Cohort B: Dose B single dose (Experimental): A single dose of GH002 or placebo administered by i.v. bolus injection (randomized as 6 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Cohort C: Dose C single dose (Experimental): A single dose of GH002 or placebo administered by i.v. bolus injection (randomized as 6 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Cohort D: Dose D single dose (Experimental): A single dose of GH002 or placebo administered by i.v. bolus injection (randomized as 6 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Cohort E: Dose E single dose (Experimental): A single dose of GH002 or placebo administered by i.v. bolus injection (randomized as 6 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Cohort F: Dose F single dose (Experimental): A single dose of GH002 or placebo administered by i.v. bolus injection (randomized as 6 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Cohort G: Dose G single dose (Experimental): A single dose of GH002 or placebo administered by i.v. bolus injection (randomized as 6 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Cohort J: Individualized Dosing Regimen (Experimental): Administration of up to 3 doses of GH002 within a single day (doses to be confirmed following review of data from single-dose part)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine

INTERVENTIONS:
Drug: 5 Methoxy N,N Dimethyltryptamine — GH002 administered via i.v. bolus injection(s)
  Other Names: GH002; 5-MeO-DMT
Drug: Placebo — GH002 placebo administered via i.v. bolus injection
  Other Names: GH002 placebo
  Arms: Cohort A: Dose A single dose; Cohort B: Dose B single dose; Cohort C: Dose C single dose; Cohort D: Dose D single dose; Cohort E: Dose E single dose; Cohort F: Dose F single dose; Cohort G: Dose G single dose

SUMMARY:
The primary objectives of this study are to investigate the safety and serum pharmacokinetics of 5-MeO-DMT in healthy volunteers in a double-blind, placebo-controlled, randomized study design with single, injected doses of GH002 and in an open-label, non-randomized study design with intra-subject dose-escalation of GH002. As secondary objectives, the PK/ pharmacodynamic relationship, PD profile of GH002 as evaluated by its psychoactive effects and impact on cognitive performance, and the serum PK of the metabolite bufotenine are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) in the range of 18.5 and 35 kg/m2 (inclusive) at Screening.
* Is deemed in good physical health by the investigator.
* Is in good mental health in the opinion of the investigator and clinical psychologist

Exclusion Criteria:

* Has known allergies or hypersensitivity or any other contra-indication to 5-MeO-DMT.
* Has received any investigational medication, including investigational vaccines, within the 6 weeks prior to baseline
* Has a current or past clinically significant condition, which renders the subject unsuitable for the trial according to the Investigator's judgement.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: incidence of treatment emergent adverse events | Up to 7 days
  Adverse events reported in the study and coded by MedDRA.
Safety and tolerability: local tolerance (injection site reactions) | Up to discharge on dosing day
  Local infusion site findings will be assessed as none, mild, moderate and severe for the following signs and symptoms of the applicable site: dryness, redness, swelling, pain, tenderness, and itching and other.
Safety and tolerability: Clinically significant changes from baseline in ECG, vital signs and safety laboratory assessments | Up to 7 days
  Clinically significant changes in ECG include any significant change in rate or rhythm as determined by the principal investigator
Safety and tolerability: Assessment of sedation (Modified Observer's Assessment of Alertness and Sedation [MOAA/S]) following each dose and as part of the discharge evaluation on Day 0 | Up to discharge on dosing day
  The Modified Observer's Assessment of Alertness and Sedation scale (MOAA/S) will be completed before and after GH002 dosing. Scored from 0 (deep sedation) to 5 (alert)
Safety and tolerability: Change from baseline in Clinician Administered Dissociative States Scale (CADSS) | Up to 7 days
  The CADSS comprises 19 subjective items, ranging from 0 'not at all' to 4 'extremely. Summed together, these subscales form a total dissociative score. Combined score ranges from 0 to 76
Safety and tolerability: Assessment of subject-discharge readiness at discharge on Day 0 | Up to discharge on dosing day
  Assessment of Discharge Readiness on the administration day by the Principal Investigator, using the Clinical Assessment of Discharge Readiness (CADR).
Safety and tolerability: Columbia-Suicide Severity Rating Scale (C-SSRS) categorization based on the Columbia Classification Algorithm of Suicide Assessment (C-CASA). | Up to 7 days
  A detailed questionnaire assessing both suicidal behaviour and suicidal ideation.
Safety and tolerability: Change from baseline in Brief Psychiatric Rating Scale (BPRS). | Up to 7 days
  A scale to measure psychiatric symptoms. Each symptom is rated 1-7 and a total of 18 symptoms are scored. Combined score ranges from 18 to 126.
The pharmacokinetic (PK) parameters derived from laboratory assay results of the systemic levels of 5-MeO-DMT | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH002 to determine 5-MeO-DMT serum concentrations.

SECONDARY OUTCOMES:
Pharmacodynamic assessment: The dose-related psychoactive effects of GH002 as evaluated by a Visual Analogue Scale | Up to 1 hour after dosing
  The Peak Experience Scale (PES) is a Visual Analogue Scale scored from 0-100
Pharmacodynamic assessment: Challenging Experiences Questionnaire (CEQ) | Up to 1 hour after dosing
  Completed by the subject after GH002 administration and assesses seven factors (grief, fear, death, insanity, isolation, physical distress, and paranoia) all scored from 0 to 5.
Pharmacodynamic assessment: 30-Question Mystical Experience Questionnaire (MEQ30) | Up to 1 hour after dosing
  The MEQ30 is a validated procedure for assessing the extent of the psychoactive effects experienced by a subject. The validated MEQ30 uses thirty assessment questions across four areas of experience, all scored from 0 to 5.
Pharmacodynamic assessment: Duration of the psychoactive effects (PsE) | Up to 1 hour after dosing
  The duration of the experience, defined as time in minutes from drug administration to time when the subject reports that any psychoactive symptoms have subsided will be recorded.
PK/PD relationship(s) of 5-MeO-DMT | Up to 1 hour after dosing
  In particular the correlation between Cmax and AUC with PES score and duration of PsE as scored by the investigator will be described
Cognitive Function: Change from baseline in Rapid visual information processing (RVP) test | Up to 7 days
  A computerized test assessing the reaction time in response to a visual stimulus.
Cognitive Function: Change from baseline in Verbal recognition memory (VRM) test | Up to 7 days
  The VRM test is based on successive auditory presentations of 18-word lists followed by attempted recall.
Cognitive Function: Change from baseline in Spatial Working Memory (SWM) task | Up to 7 days
  The SWM test requires retention and manipulation of visuospatial information. This test has notable executive function demands, and measures strategy use as well as errors. In this task the subject has to search for tokens hidden in boxes on screen. The subject must touch a box to open the box to reveal either a yellow token or an empty box. Once the subject has found a yellow token, they must touch the outline of the right-hand side of the screen to 'store' it. The subject must then continue searching through the boxes until all of the tokens have been found. The test takes about 4 minutes to complete
Cognitive Function: Change from baseline in Digit Symbol Substitution Task (DSST) | Up to 7 days
  The DSST is a global measure of cognitive ability, requiring the engagement of multiple cognitive domains in order to complete effectively. A computerized test with the task is to match digits with symbols from encoding list. The number of digits correctly encoded within 90 seconds is the performance measure.
The pharmacokinetic (PK) parameters derived from laboratory assay results of the systemic levels of bufotenine | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH002 to determine bufotenine serum concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- GH Research Clinical Trial Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No